CLINICAL TRIAL: NCT06214416
Title: Pragmatic Clinical Trial to Compare the Short and Medium Term Effects of Two Recommendations Regarding Alcohol Consumption: a Pilot Study NAMETI_ALCOHOL
Brief Title: Pragmatic Clinical Trial of Two Recommendations Regarding Alcohol Consumption: a Pilot Study NAMETI_ALCOHOL
Acronym: NAMETI_ALCOHOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Ministry of Health, Spain (Other Government)
Responsible Party: Principal Investigator, Maira Bes Rastrollo, Professor, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NAMETI_ALCOHOL_10_2020
Record Dates: First submitted 2022-05-25; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: It is intended to recruit a total of 100 participants, including two observational cohorts of abstainers and drinkers. The intervention will be carried out in drinkers willing to change their alcohol consumption, divided into 2 groups of 150 participants, the abstention group and the Mediterranean alcohol-drinking pattern group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Abstention (Active Comparator): These participants will be encouraged to totally avoid alcohol consumption.
  Interventions: Behavioral: Abstention
- Mediterranean alcohol-drinking pattern (Active Comparator): These participants will be encouraged to change their pattern of consumption to a more Mediterranean way, which includes 5 aspects: moderate alcohol consumption (maximum of 2 drinks/day for women and 4 drinks/day for men), spread consumption throughout the week, drink with meals and never with an empty stomach, prefer wine and mainly red wine, as well as completely avoid episodes of binge-drinking.
  Interventions: Behavioral: Mediterranean alcohol-drinking pattern
- Control of abstainers (No Intervention): This group will include all participants who consume less than 3 alcohol drinks a week at the time of recruitment.
- Control of drinkers (No Intervention): This group will include all participants who don't want to change their alcohol-drinking pattern.

INTERVENTIONS:
Behavioral: Abstention — All the intervention will be carried out online once a month for a year, focusing on nutritional, behavioral and scientific evidence aspects, that promote abstention.
  Arms: Abstention
Behavioral: Mediterranean alcohol-drinking pattern — All the intervention will be carried out online once a month for a year, focusing on nutritional, behavioral and scientific evidence aspects, that promote the Mediterranean alcohol-drinking pattern.
  Arms: Mediterranean alcohol-drinking pattern

SUMMARY:
NAMETI-Alcohol, from the acronym for Navarra Medical Trialist Initiative, is a pilot study in which two patterns of alcohol consumption, abstention and Mediterranean alcohol-drinking pattern, and their effects on health in the short and medium term will be compared.

DETAILED DESCRIPTION:
Background: Alcohol is the most consumed psychoactive substance in Spain. In 2016 it was the seventh leading risk factor for death and disability-adjusted lost years worldwide, and the first one in people between 15 and 49 years old.In the scientific community there is some controversy about what would be the best approach to face this great problem. On the one hand, there is evidence to recommend that there is no safe level of alcohol. However, on the other hand, there are studies that demonstrate the protective role of a moderate alcohol consumption. In this pilot study both options will be compared.

Methods: It is intended to recruit a total of 100 participants, including two observational cohorts of abstainers and drinkers. The intervention will be carried out in drinkers willing to change their alcohol consumption, divided into 2 groups of 50 participants, the abstention group and the Mediterranean alcohol-drinking pattern group. The Mediterranean alcohol-drinking pattern includes 5 aspects: moderate alcohol consumption (maximum of 1 drinks/day for women and 2 drinks/day for men), spread consumption throughout the week, drink with meals and never with an empty stomach, prefer wine and mainly red wine, as well as completely avoid episodes of binge-drinking. The main objective will be to compare the short and medium term effects on health of both patterns.

ELIGIBILITY:
Inclusion Criteria:

* Consuming more than 3 drinks a week (except for the abstention-control arm)

Exclusion Criteria:

* Sever chronic disease (cancer, cardiovascular disease, chronic hepatitis and mental illness)
* Pregnant women or breastfeeding
* Family or personal history of addiction, alcoholism or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Glucose (mg/dl) | 1 year
  Changes differences in glucose levels
HDL-Cholesterol (mg/dl) | 1year
  Changes differences in HDL-Cholesterol levels
Total cholesterol (mg/dl) | 1year
  Changes differences in total cholesterol levels
Triglycerides (mg/dl) | 1 year
  Changes differences in triglycerides
Alanine Aminotransferase (ALT) (IU/L) | 1 year
  Changes differences in ALT
Aspartate transaminase (AST) (IU/L) | 1 year
  Changes differences in AST
Gamma-glutamyltransferase (GGT) (IU/L) | 1 year
  Changes differences in GGT
c-Reactive Protein (CRP) (mg/L) | 1 year
  Changes differences in CRP
Blood pressure (mm Hg) | 1 year
  Changes differences in systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Mental health | 1 year
  Through Beck's questionnaire, Lobo's mini-cognitive exam (Mini-Mental State examination) and clock drawing test
Weight (kg) | 1 year
  Changes in weight (kg)
Adherence to the intervention | 1 year
  Levels of resveratrol in urine and hydroxytyrosol in plasma and urine
Body Mass Index (BMI) (kg/m2) | 1 year
  Changes in BMI, assessed through weight(kg) and height (m) (BMI=Weight/(Height)^2

CONTACTS AND LOCATIONS:
Locations (1):
- University of Navarra, Pamplona, Navarre, Spain